CLINICAL TRIAL: NCT02038153
Title: A Phase I/II Study of Lenalidomide Maintenance After Autologous Stem Cell Transplant for Elderly Patients With Acute Myeloid Leukemia (AML)
Brief Title: Lenalidomide in Treating Older Patients With Acute Myeloid Leukemia Who Have Undergone Stem Cell Transplant
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ira Braunschweig, Principal Investigator, Albert Einstein College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-08-148; NCI-2013-02493 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13-08-148 (Other: Albert Einstein College of Medicine); P30CA013330 (NIH)
Record Dates: First submitted 2014-01-15; First posted 2014-01-16 (Estimated); Results first posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Adult Acute Myeloid Leukemia in Remission
MeSH Terms: interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (lenalidomide) (Experimental): Patients receive lenalidomide PO QD on days 1-21. Courses repeat 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Lenalidomide

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid

SUMMARY:
This phase I/II trial studies the side effects and best dose of lenalidomide and how well it works in treating older patients with acute myeloid leukemia (AML) who have undergone stem cell transplant. Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and efficacy of maintenance lenalidomide post autologous peripheral blood stem cell transplantation (PBSCT) for elderly patients with AML (AML).

SECONDARY OBJECTIVES:

I. To define maximum tolerated dose (MTD) and establish therapeutic dose level (TDL) of lenalidomide given post autologous transplant for AML.

II. To determine the progression free survival for patients treated with this approach.

III. To determine the overall survival for patients treated with this approach. IV. To determine the role of residual AML stem cells on efficacy of lenalidomide maintenance after autologous PBSCT.

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

Patients receive lenalidomide orally (PO) once daily (QD) on days 1-21. Courses repeat 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed diagnosis of non-M3 AML; antecedent myelodysplastic syndrome (MDS) is acceptable
* Post autologous stem cell transplant bone marrow biopsy core that is consistent with morphologic remission
* Must have received induction and consolidation chemotherapy, and autologous stem cell transplant for AML
* Life expectancy of greater than 12 months
* Karnofsky performance status 70 or greater
* Leukocytes >= 2,000/mcL
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 75,000/mcL
* Total bilirubin =< 4 X institutional upper limit of normal unless 2nd to Gilbert's disease
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 4 X institutional upper limit of normal
* Creatinine < 1.5 X institutional upper limit of normal OR creatinine clearance >= 30 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Able to take aspirin, or warfarin, or low molecular weight heparin as prophylactic anticoagulation
* Ability to understand and the willingness to sign a written informed consent document
* Must be registered into the mandatory RevAssist® program and be willing and able to comply with the requirement of RevAssist®

Exclusion Criteria:

* Patient received chemotherapy or radiotherapy within 2 weeks prior to entering the study or has not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patient received another investigational agent after post autologous stem cell transplant
* Patient who will be receiving another investigational product during the study
* Patient who is growth factor or transfusion dependent
* Patient has central nervous system leukemia
* History of allergic reactions attributed to thalidomide or lenalidomide
* History of erythema nodosum, characterized by a desquamating rash while taking thalidomide or similar drugs
* Prior history of metastatic malignancy
* Uncontrolled illness including, but not limited to ongoing or active infection, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; patients must not have suffered recent (< 6 months) myocardial infarction, unstable angina, uncontrolled hypertension, or difficult to control cardiac arrhythmias
* Evidence of uncontrolled congestive heart failure
* Active hepatitis B as defined by hepatitis B surface antigen positivity, unless able to start dual anti-hepatitis B (HepB) therapy, or already on dual anti-HepB therapy
* Patients who are positive for hepatitis B core antibody, but negative for the hepatitis B surface antigen, should be on lamivudine 100 mg daily until at least 3 months post-transplant
* Patient is positive for human immunodeficiency virus (HIV) or human T-cell lymphotropic virus-1 (HTLV-1)
* Women of childbearing potential (defined as a sexually mature woman who has not undergone a hysterectomy or who has had menses at any time in the preceding 24 consecutive months)
* Men who did not agree not to father a child and who refused to use a latex condom during any sexual contact with women of childbearing potential while taking lenalidomide and for 4 weeks after therapy is stopped, even if they have undergone a successful vasectomy

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-12; Primary Completion 2015-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ira Braunschweig, Principal Investigator — Albert Einstein College of Medicine
Locations (3):
- United States (3):
  - Albert Einstein College of Medicine, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Lenalidomide)
Started | 3
Completed | 2
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Lenalidomide)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 2
  Hispanic | 1
  White | 0
  Asian | 0

OUTCOME MEASURES:

1. Primary Outcome: Relapse Free Survival Rate
Description: The Relapse free survival rate is defined as the Leukemia free survival rate during the first two years after and during the initiation of treatment . The observed relapse free survival rate will be calculated along with its 95% confidence interval. A one sample test on proportion will be used to detect if the relapse free survival rate with lenalidomide is significantly higher than that without the treatment (relapse rate is expected to be > 95%).
Time Frame: initial 2 years after treatment begins
Population: Study terminated because of low accrual. No analysis done
Arm/Group | Treatment (Lenalidomide)
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Survival
Description: Kaplan-Meier analysis will be conducted.
Time Frame: From transplant until death of any cause, assessed up to 5 years
Population: Study terminated because of low accrual. No analysis done
Arm/Group | Treatment (Lenalidomide)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Treatment (Lenalidomide)
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-01-03): https://cdn.clinicaltrials.gov/large-docs/53/NCT02038153/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT02038153/ICF_001.pdf